CLINICAL TRIAL: NCT06569199
Title: Functional Bracing Versus Spica Casting for the Treatment of Pediatric Diaphyseal Femur Fractures: A Randomized Prospective Study and Cost-effectiveness Analysis
Brief Title: Pediatric Femur Fractures: Functional Bracing vs Spica Casting - Outcomes and Cost Analysis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: OrthoPediatrics (2850 Frontier Drive Warsaw, IN, USA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB24-0318
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-04

CONDITIONS: Pediatric Femur Fracture
Keywords: Functional Brace; Hip Spica Cast; Orthopedic Surgery; Pediatric

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants and parents are blinded until after study has been explained and consent obtained. Participants then are randomized into either the spica cast or functional bracing group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Bracing (Experimental): Premade fabricated braces in three sizes (small, medium and large) that have been designed for the pediatric age group between 0-5 years old will be stocked at the Alberta Children's Hospital. Participants who are randomized to the functional bracing group will be administered the functional brace within the emergency department under light procedural sedation. Brace will be used for up to 8 weeks administration until adequate callous formation confirmed with X-ray imaging.
  Interventions: Device: Functional Bracing
- Hip Spica Cast (Active Comparator): Participants who are randomized to the spica casting group will undergo casting in the operating room and be given general anesthesia to apply the hip spica cast. Cast will be used for up to 8 weeks administration until adequate callous formation confirmed with X-ray imaging.
  Interventions: Device: Hip Spica Cast

INTERVENTIONS:
Device: Functional Bracing — Premade fabricated braces in three sizes (small, medium and large) that have been designed for the pediatric age group between 0-5 years old will be stocked at the Alberta Children's Hospital. Braces will be applied to participants in the emergency department. As these braces are designed to allow for positional adjustments, if deemed necessary adjustments will be made by the attending orthopaedic surgeon at subsequent follow-up visit(s).
  Arms: Functional Bracing
Device: Hip Spica Cast — The current standard of care for diaphyseal pediatric hip fractures in children aged 6 months to 5 years old is hip spica casting. A hip spica is a hard cast that covers a child's body from the chest down to their knees or ankles allowing for fracture immobilization to promote healing. Application of the spica cast occurs in the operating room and requires a general anaesthetic. Caring for a child in a hip spica cast presents significant challenges for caregivers due to the cast's cumbersome size and restricted mobility which makes routine caregiver activities like daily hygiene, toileting, transportation and skin surveillance difficult. Inadequate maintenance of the spica cast may result in skin complications, necessitating extra visits for cast adjustments, or potentially requiring revision casting in the operating room.
  Arms: Hip Spica Cast

SUMMARY:
Pediatric diaphyseal femur fractures that occur in children aged 6 months to 5 years old are traditionally treated with hip spica casting. However, recent studies suggest that functional bracing may offer clinical and financial benefits, yet there's a lack of prospective trials comparing these two treatment methods. This single-center randomized-control trial aims to assess subjective and objective clinical outcomes as well as financial aspects of functional bracing versus spica casting. Functional bracing, proposed as a potentially superior alternative, may address caregiver challenges and reduce costs by avoiding operating room time and hospital admissions. The study will evaluate fracture reduction, time to union, functional outcomes, and caregiver satisfaction. Additionally, a comprehensive cost-effectiveness analysis will be conducted. Ultimately, this research aims to inform clinical decision-making regarding the optimal management of pediatric femur fractures, considering both clinical effectiveness and economic implications.

DETAILED DESCRIPTION:
Pediatric diaphyseal femur fractures are a common orthopedic injury in children, with about one-third occurring in patients under the age of five. These fractures require effective management to promote optimal healing and functional recovery. In the 6-month to 5-year-old age group, diaphyseal femur fractures have traditionally been treated with a hip spica cast. Application of a hip spica cast typically occurs in the operating room (OR) under general anesthesia given that patients must undergo prolonged sedation for cast application. Caring for a child with a hip spica cast presents significant challenges for caregivers due to the cast's cumbersome size and restricted mobility. This makes routine activities such as daily hygiene, toileting and skin surveillance difficult for caregivers. An ecological study performed by Kocher et al. found that spica casting places a greater burden on family functioning than medical treatment in children with serious chronic medical conditions including diabetes, renal failure, and juvenile rheumatoid arthritis.1

Kramer et al. have recently proposed the use of functional bracing as an equally effective alternative to traditional hip spica casting for the treatment of pediatric diaphyseal femur fractures. In their study, they found no differences in the correction and maintenance of fracture alignment, time to union and functional outcomes2. The use of a prefabricated and adjustable functional brace was suggested to be better tolerated by patients and their parents as the open design allows for improved hygiene, ease of cleaning, toileting, skin surveillance and improved positional movement.

From a cost-effectiveness analysis perspective, it has been inferred that the overall cost of functional bracing compared to spica casting is lower as it can be applied in the emergency department without the need for a general anesthetic or operating room time. Furthermore, we hypothesize that functional bracing will also decrease visits to orthopedic clinics for cast-related issues which will further decrease the overall costs associated with the treatment of pediatric diaphyseal fractures with a functional brace when compared to a hip spica cast. Having said this, no comprehensive cost-effectiveness analysis studies have been performed to our knowledge and there is minimal literature comparing functional bracing versus spica casting for the treatment of pediatric diaphyseal femur fractures.

This proposed study aims to address this gap by conducting a randomized prospective study comparing functional bracing and spica casting for the treatment of pediatric diaphyseal femur fractures by evaluating maintenance of fracture reduction, time to union, leg-length, functional outcomes, complications, parent/caregiver satisfaction with the treatment as well as performing a supplemental comprehensive cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 6mo-5 years
* Isolated closed diaphyseal femur fracture
* Parent or caregiver 18 years of age or older who are cognitively able to complete the parent/caregiver satisfaction survey.

Exclusion Criteria:

* Patients <6 months or >5 years of age
* Underlying neuromuscular disorders
* Open diaphyseal femur fracture
* Polytrauma
* Medical comorbidities impacting fracture healing
* <6 week follow-up

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Time to union/rate of non-union | Post-intervention clinical follow-ups up to 1 year
  Assessed by radiographic evidence at clinic follow-up visits.
  This will be measuring the length of time and changes in union of bone, and to see if the bone has not healed properly.
Rates of malunion | Post-intervention clinical follow-ups up to 1 year
  Assessed by radiographic evidence at clinic follow-up visits.
  Malunion defined as 6 months-2years: > 30 degrees varus/valgus; >30 degrees procurvatum; or >15 mm shortening.
  2 years-5 years: > 15 degrees varus/valgus; > 20 degrees procurvatum; or >20 mm shortening.
Changes in Leg Length | Post-intervention clinical follow-ups up to 1 year
  Assessed by radiographic evidence at clinic follow-up visits.
  Leg length will be measured using radiographs to determine if there any changes to leg length or discrepancies compared to the contralateral side.
Flynn Score | 6 weeks post intervention and at 1 year post-intervention
  Flynn Scoring system will be used to determine final functional results. The Flynn scoring system classifies functional results as: excellent, satisfactory or poor. An excellent result is defined as leg-length discrepancy <1.0cm, femoral malalignment <5 degrees, no pain and no complications. Satisfactory result is defined as leg-length discrepancy <2.0cm, femoral malalignment 5-10 degrees, no pain as well as minor and resolved complications. A poor result is defined as leg-length discrepancy >2.0cm, femoral malalignment >10 degrees, presence of pain and major and lasting complications. Flynn score will be calculated at the 6 week mark and 1 year mark.
Number of radiographs and cast clinic visits | Post-intervention clinical follow-ups up to 1 year
  This will be used to determine which arm had less radiation from radiographs and less visits with the surgeon.
Pediatric Outcome Data Collection Instrument (PODCI) | Post-intervention clinical follow-ups up to 1 year
  a validated patient-reported quality of life and outcome measure primarily used to assess motor function following orthopedic surgical intervention. Will be completed by the parent at the 6-week and 1-year post-intervention visit and will allow for us to determine subjective outcomes.
Complications | Post-intervention clinical follow-ups up to 1 year
  Includes skin break down issues, pressure sores, repeat operative intervention, cast or brace related issues.
Parent Satisfaction Survey | At 6 week and 1 year follow-up.
  The caregiver will complete both the Impact on Family Scales (IFS) and EQ-5D questionnaires. The IFS is a validated 27-item score with Likert-scaling that measures the impact of children's health conditions on his/her family life that addresses four domains: economic impact on family, social impact, familial impact and personal strain/coping. The EQ-5D questionnaire is a brief validated questionnaire designed to evaluate mobility, self-care, usual activities, pain and discomfort as well as anxiety and depression.
Economic costs | Initial presentation to hospital up to 1 year
  Direct costs associated with treatment, including materials, equipment, and hospital stays, OR costs, emergency room visit costs will be compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Phillips, MD, Principal Investigator — University of Calgary; David Parsons, MD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen V, Sanders JS, Skaggs DL, Kay RM, Andras LM. (2022). Functional Bracing of Femur Fractures in Young Children Avoids Anesthesia and Spica Casting with Equivalent Outcomes: A Randomized Prospective Study: 2022 POSNA Annual Meeting. Journal of the Pediatric Orthopaedic Society of North America, 4(3).
- [Background] Kramer AS, JS, Woon C, Speers D, (2016). Functional Bracing for Treatment of Pediatric Diaphyseal Femur Fractures: An Alternative to Spica Casting: 2016 POSNA Annual Meeting. Journal of the Pediatric Orthopaedic Society of North America.
- [Background] Kocher, M., Ciarlo, M., Feroe, A., Dichtel, L., & Traver, J. (2022). Impact on Family Functioning of Immediate Spica Casting for Pediatric Femur Fractures: An Ecological Study: Original Research. Journal of the Pediatric Orthopaedic Society of North America, 4(1).
- [Background] Rockwood C.A., Beaty J.H., Kasser J.R. Lippincott Williams & Wilkins; 2010. Rockwood and Wilkins' Fractures in Children.
- [Background] Flynn JM, Luedtke LM, Ganley TJ, Dawson J, Davidson RS, Dormans JP, Ecker ML, Gregg JR, Horn BD, Drummond DS. Comparison of titanium elastic nails with traction and a spica cast to treat femoral fractures in children. J Bone Joint Surg Am. 2004 Apr;86(4):770-7. doi: 10.2106/00004623-200404000-00015. PMID 15069142